CLINICAL TRIAL: NCT07147582
Title: Effect of Transcranial Alternating Current Stimulation on Sleep Disorder and Anxiety in Elderly Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salah Eid Ahmed Ali, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SREC.PT.SUE(14)625
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Sleep Disorders; Anxiety Disorder
Keywords: Anxiety; Elderly; Sleep Dsorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Transcranial alternating current stimulation activating brain alpha wave
  Interventions: Other: Transcranial alternating current stimulation with two electrodes placed on scalp
- control (Sham Comparator): Transcranial alternating current stimulation will not be turned on
  Interventions: Other: Transcranial alternating current stimulation with two electrodes placed on scalp

INTERVENTIONS:
Other: Transcranial alternating current stimulation with two electrodes placed on scalp — Transcranial alternating current stimulation with anode and cathode electrodes and frequency ranged from 8 to 13 HZ

SUMMARY:
Sleep disorders and anxiety are complicated disorders affecting population especially elderly population, therefore treating these disorders will have positive impact on population production and quality of life.

DETAILED DESCRIPTION:
Alternating current cranial stimulation will improve brain waves frequency so that will have positive effect on sleep disorders and anxiety on elderly population.

ELIGIBILITY:
Inclusion Criteria:

-healthy elderly adult aged more than 60 years old, both sex, and suffering from insomnia and sleep disorders

Exclusion Criteria:

* neurological and vascular diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | before treatment and after 12 weeks
  Pittsburgh Sleep Quality Index (PSQI) will be used for sleep quality assessment Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties

SECONDARY OUTCOMES:
Anxiety | before treatment and after 12 weeks of treatment
  Hamilton's Depression Scale (HAMA) will be used to assess level of anxiety rated from 0 to 4 with 0 represent absent and 4 represent more severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No